CLINICAL TRIAL: NCT02990858
Title: An Extension Protocol for Subjects Who Successfully Completed PRO140_CD02 or PRO140_CD02_Open Label Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA required the sponsor to halt enrollment in the trial and transition participants to available therapies for the treatment of their disease. The trial was subsequently terminated once participants were transitioned.
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140 _CD02 Extension
Record Dates: First submitted 2016-11-17; First posted 2016-12-13 (Estimated); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leronlimab (PRO 140) (Experimental): The treatment extension phase consists of weekly treatment injection of PRO 140 in addition to Optimized Background Therapy.
  Interventions: Drug: PRO 140

INTERVENTIONS:
Drug: PRO 140 — PRO 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5). Participants received 350 or 700 mg weekly injections of PRO 140.
  Other Names: Leronlimab

SUMMARY:
PRO 140_CD02 Extension study seeks to evaluate the long-term efficacy, safety and tolerability of PRO 140 weekly injection in combination with Optimized Background Therapy (OBT) in patients infected with Human Immunodeficiency virus (HIV-1).

DETAILED DESCRIPTION:
This is an extension study, to provide continued access to PRO 140 to subjects who complete participation in PRO140_CD02 and continue to receive clinical benefit and would require PRO 140 to form a viable regimen, in the opinion of the treating physician. The patient population for this trial are treatment-experienced HIV infected patients with C-C Chemokine Receptor Type 5 (CCR5)-tropic virus who demonstrate evidence of HIV-1 suppression after successfully completed 24 weeks of treatment in the PRO140_CD02 or CD02_OpenLabel study.

ELIGIBILITY:
Inclusion Criteria: Potential subjects are required to meet all of the following criteria for enrollment into the study.

1. Subjects who have completed 24 weeks of treatment in PRO 140_CD 02 or CD02_OpenLabel study, and Investigator believes subject requires continued access to PRO 140 in order to continue deriving clinical benefit and maintain HIV-1 viral suppression.
2. HIV-1 RNA ≤ 50 copies/ml at T23 Visit in PRO140_CD02 study
3. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized).

   Females of childbearing potential must have a negative urine pregnancy test prior to receiving the first dose of study drug.
4. Willing and able to participate in all aspects of the study, including use of subcutaneous (SC) medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria: Potential subjects meeting any of the following criteria will be excluded from enrollment.

1. Not currently enrolled in PRO 140_CD 02 or CD02_OpenLabel study
2. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma)
3. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
4. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Principal Investigator — CytoDyn, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 43 participants in the United States.
Groups:
- PRO 140: Eligible subjects received 350 mg or 700 mg PRO 140 (leronlimab) administered weekly as subcutaneous injections along with Optimized Background Therapy (OBT) until virologic failure or another reason for discontinuation.
Period: Overall Study
Arm/Group | PRO 140
Started | 43
Completed | 23
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Arm/Group | PRO 140
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.07 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Viral Load (HIV-1 RNA Levels) at the Conclusion of Treatment Period
Description: The change from baseline in HIV-1 RNA levels (log 10 copies/mL) was summarized at least once every four weeks during the treatment extension phase. The time-weighted mean of change of the post baseline values was calculated. The time-weighted mean was adjusted AUC (area under the curve) by time.
Time Frame: From TE1 (first treatment administration) to once every four weeks until last treatment visit (up to 56 months).
Population: The analysis population is defined as all subjects who enrolled in the study and received at least one dose of PRO 140. Subjects who had undefined change from baseline due to missing data were excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | PRO 140
Number analyzed (Participants) | 43
log10 copies/mL | 0.13 (1.11)

2. Secondary Outcome: Mean Change in CD4 Cell Count at the Conclusion of Treatment Period
Description: The change from baseline in CD4 cell count was summarized for each visit during the treatment phase. The time-weighted mean of change of the post baseline values was calculated. The time-weighted mean was adjusted AUC (area under the curve) by time.
Time Frame: From first treatment administration to each weekly visit until the last treatment visit (up to 56 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | PRO 140
Number analyzed (Participants) | 43
cells/uL | 46 (122)

3. Secondary Outcome: Proportion of Participants Experiencing Emergence of Dual/Mixed (D/M)- and CXCR4-tropic Virus in Patients Who Had Exclusive CCR5-tropic Virus at Study Entry.
Description: All patients have exclusive C-C chemokine receptor type 5 (CCR5)-tropic virus at study entry. The proportion of patients with any tropism result of dual/mixed was summarized.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 56 months.
Population: The analysis population is defined as all subjects who enrolled in the extension portion of the study and received at least one dose of PRO140. Participants who had no dual/mixed tropism data collected or had undefined change from baseline due to missing data were excluded from the analysis.
Measure: Number; unit: proportion of participants
Arm/Group | PRO 140
Number analyzed (Participants) | 37
proportion of participants | 0.093

4. Secondary Outcome: Tolerability of Repeated Subcutaneous Administration of PRO 140 as Assessed by Investigator Evaluation of Injection Site Reactions (ISR)
Description: At each visit during the treatment extension phase, an injection site reaction assessment was completed for the current and previous injection sites. To assess severity, subcutaneous (SC) injection related events were recorded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table).
  Grade 1 indicates a mild event Grade 2 indicates a moderate event Grade 3 indicates a severe event Grade 4 indicates a potentially life-threatening event Participants who had no symptoms of injection site reactions, "0" was assigned.
Time Frame: From TE1 (first treatment administration) weekly until last treatment visit (up to 56 months).
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population. Subjects who had undefined value due to missing data were excluded from the analysis population.
Measure: Number; unit: participants
Arm/Group | PRO 140
Number analyzed (Participants) | 39
participants
  Participants with no ISR symptoms | 20
  Participants with Grade 1 ISR | 19
  Participants with Grade 2 or higher ISR | 0

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events Resulting in Study Drug Discontinuation
Description: Treatment-related adverse events are defined as events with an onset on or after the first treatment (TE1).
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 56 months.
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Measure: Number; unit: participants
Groups:
- PRO 140: Eligible subjects received either 350 mg or 700 mg PRO 140 (leronlimab) administered weekly as subcutaneous injections along with Optimized Background Therapy (OBT) until virologic failure or another reason for discontinuation.
Arm/Group | PRO 140
Number analyzed (Participants) | 43
participants | 1

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events as Defined by the DAIDS Adverse Event Scale
Description: The Division of AIDS (DAIDS) grading table provides an adverse event severity grading scale ranging from grades 1 to 5 with descriptions for each adverse event based on the following general guidelines:
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death (Note: This grade is not specifically listed on each page of the grading table).
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 56 months.
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Measure: Number; unit: participants
Arm/Group | PRO 140
Number analyzed (Participants) | 43
participants | 12

7. Secondary Outcome: Number of Participants With at Least One Treatment-related Serious Adverse Event.
Description: Treatment-related (as defined by the investigator) serious adverse events are defined as serious events with an onset on or after the first treatment.
  A serious adverse event is defined as any adverse event that:
  * Results in death
  * Is life threatening (the subject is at immediate risk of dying from the AE)
  * Requires subject hospitalization or prolongs existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 56 months.
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140
Number analyzed (Participants) | 43
Participants | 15

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the first treatment extension visit and continue up until the final study visit, up to 56 months.
Description: Adverse events were elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the Investigator believed were clinically significant to the research subject and that occurred after initiation of the first study treatment was reported as an adverse event.
Groups:
- PRO 140 350 mg: Eligible subjects received 350 mg PRO 140 (leronlimab) administered weekly as subcutaneous injections along with Optimized Background Therapy (OBT) until virologic failure or another reason for discontinuation.
- PRO 140 700 mg: Eligible subjects received 700 mg PRO 140 (leronlimab) administered weekly as subcutaneous injections along with Optimized Background Therapy (OBT) until virologic failure or another reason for discontinuation.
Arm/Group | PRO 140 350 mg | PRO 140 700 mg
All-Cause Mortality (participants affected / at risk) | 3/29 | 1/14
Serious Adverse Events (participants affected / at risk) | 11/29 | 4/14
Other Adverse Events (participants affected / at risk) | 27/29 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 350 mg (N=29) | PRO 140 700 mg (N=14)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 350 mg (N=29) | PRO 140 700 mg (N=14)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (10) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 2 (6)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 5 (10) | 1 (1)
Chest pain (General disorders) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Sinusitis (Infections and infestations) | 4 (6) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 2 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (7)
Abdominal rebound tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood HIV RNA increased (Investigations) | 0 (0) | 1 (6)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lip Injury (Investigations) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Renal and urinary disorders) | 3 (3) | 0 (0)
Red blood cells urine (Investigations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Scapula pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Olecranon bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
FDA required the sponsor to halt enrollment in the trial and transition participants to available therapies for the treatment of their disease. The trial was subsequently terminated once participants were transitioned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT02990858/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT02990858/SAP_001.pdf